CLINICAL TRIAL: NCT03808103
Title: A Phase 1/2a Double-Blind, Randomized, Placebo-Controlled Trial to Assess the Safety and Efficacy of Oral Administration of EcoActive on Intestinal Adherent Invasive Escherichia Coli (AIEC) in Patients With Inactive Crohn's Disease (CD)
Brief Title: Safety and Efficacy of EcoActive on Intestinal Adherent Invasive E. Coli in Patients With Inactive Crohn's Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intralytix, Inc. (Industry)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITX/EA-002
Record Dates: First submitted 2019-01-04; First posted 2019-01-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
Keywords: Phage; Bacteriophage; AIEC
MeSH Terms: conditions — Crohn Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Dose is 1mL of placebo given orally twice a day for 15 days
  Interventions: Biological: Placebo
- Phage (Experimental): Dose is 1mL of bacteriophage preparation given orally twice a day for 15 days
  Interventions: Biological: Bacteriophage preparation

INTERVENTIONS:
Biological: Placebo — Orally, twice a day, for a period of fifteen days
  Other Names: 0.9% saline
  Arms: Placebo
Biological: Bacteriophage preparation — Orally, twice a day, for a period of fifteen days
  Other Names: EcoActive
  Arms: Phage

SUMMARY:
This study will evaluate the safety of oral administration of EcoActive to patients with inactive Crohn's disease and how it affects the levels of AIEC in stool.

DETAILED DESCRIPTION:
The purpose of this study is to determine if EcoActive is safe and effective in people with Crohn's disease. EcoActive is a collection of bacteriophages. Bacteriophages (or phages) are viruses that infect only bacteria. The phages in EcoActive infect a specific type of bacteria called Adherent Invasive Escherichia coli (AIEC).

The cause of Crohn's disease is poorly understood. However, the presence of AIEC in the intestines is associated with worsening inflammation in this disease. Inflammation is the presence of redness, irritation, and ulcers in the intestines. By using phages that only infect and kill this specific type of bacteria (AIEC), it is the hope this can be used to improve the course of Crohn's disease. The phages would only target the AIEC, without affecting the natural, often helpful, bacteria of the intestines. EcoActive may also lessen the use of antibiotics to control symptoms. When antibiotics are used, they can have major effects on the rest of the bacteria in the intestines. Also, repeated use can cause intestinal bacteria to become resistant to antibiotics. Reduced use of antibiotics would limit both of these risks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Inactive Crohn's disease in clinical and objective remission with a Harvey-Bradshaw Index (HBI) < 4
3. Permitted CD medications expected to remain stable during the period of the study (see Section 7 "Concomitant Crohn's Disease Medications" for allowed and prohibited drugs).
4. Crohn's disease history ≥ 6-month duration
5. CRP (C-reactive protein) within normal range at the Screening visit (based on normal range of the local laboratory)
6. Fecal calprotectin level ≤ 150 µg/g at the Screening visit
7. AIEC detected in the stool
8. Females of childbearing age must be using an effective method of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the study (contraceptive measures considered adequate are: intrauterine devices, hormonal contraceptives, such as contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release).
9. Negative pregnancy test for women of childbearing age (menarche to menopause)
10. Patient understands the study procedures, and can sign the informed consent, and the authorization to release relevant protected health information to the Study Investigator.

Exclusion Criteria:

1. Active Crohn's disease with a Harvey-Bradshaw Index (HBI) ≥ 4
2. Ongoing gastrointestinal pathology: colorectal tumor, gastrointestinal bleeding
3. Active malignancies or any malignant disease within the past 5 years
4. Indeterminate colitis, ulcerative colitis
5. Colectomy or partial colectomy (less than ileo-transverse colonic anastomosis).
6. Colonic or small bowel stoma
7. Active perianal lesions
8. Women who are pregnant or nursing, or plan to become pregnant during the study period
9. Severe uncontrolled diseases that could increase the risk for subjects participating in the study, including but not limited to: heart diseases, congestive heart failure, hypertension, lung diseases; endocrine diseases; clinically significant renal disease characterized by a glomerular filtration rate < 60mL/min, hepatic diseases, haematological disorders, or other conditions that in the opinion of the Investigator could interfere with the interpretation of the study results.
10. Taking supplemental probiotics in the form of pills or tablets.
11. History or planned procedures specifically aimed at modifying the gastrointestinal microbiota within the past year.
12. Topical gastrointestinal treatment (e.g., enemas) in the 2 weeks prior to the Screening visit or planned during the study period
13. Use of bowel cleansing or preparation for endoscopy, TDM or MRI in the 4 weeks prior to the Screening visit or planned during the study period.
14. Receipt of antibiotics 4 weeks before the Screening visit or planned during the study period.
15. Known allergy or hypersensitivity to an excipient in the study drug or placebo
16. Psychological or linguistic incapability to sign the informed consent.
17. Lack or expected lack of cooperation or compliance with the study.
18. Receipt of mesalamine based therapies within 4 weeks of the screening visit.
19. Severe psychiatric, psychological, or neurological disorders.
20. Alcohol, drug or medication abuse within the past year.
21. Subject who cannot be contacted in case of emergency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  The number of solicited and unsolicited adverse events will be recorded.
Severity of adverse events | Up to 6 months
  The severity will be graded according to the definitions and values stated in CTCAE V04 v4.
Effect on Harvey Bradshaw Index (HBI) | Up to 6 months
  The effect on Crohn's disease activity will be evaluated using the HBI.
Effect on inflammation, as indicated by C-reactive protein (CRP) | Up to 6 months
  The changes in CRP from baseline will be evaluated.
Effect on inflammation, as indicated by fecal calprotectin | Up to 6 months
  The changes in fecal calprotectin levels from baseline will be evaluated.

SECONDARY OUTCOMES:
Effect on the incidence and levels of AIEC | Up to 6 months
  The secondary objective is to assess the effect of oral phage administration on the AIEC (CFU/g) in stools of patients receiving phages vs. patients receiving placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hirten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Reezwana Chowdhury, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Green Spring Station, Lutherville, Maryland
  - Icahn School of Medicine at Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lenneman BR, Fernbach J, Loessner MJ, Lu TK, Kilcher S. Enhancing phage therapy through synthetic biology and genome engineering. Curr Opin Biotechnol. 2021 Apr;68:151-159. doi: 10.1016/j.copbio.2020.11.003. Epub 2020 Dec 10. PMID 33310655